CLINICAL TRIAL: NCT02173405
Title: Pelvic Floor Trigger Point Injection With OnabotulinumtoxinA for the Treatment of Severe Myofascial Pelvic Pain (MPP) - A Randomized, Controlled Trial
Brief Title: Injection With OnabotulinumtoxinA (Botox) for the Treatment of Chronic Pelvic Pain
Acronym: BotoxMPP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Sangetta Mahajan MD, Assistant Professor & Head Division of Female Pelvic Medicine/Reconstructive Surgery/Obstetrics/Gynecology/Urology and Director of joint fellowship in Female Pelvic Medicine andReconstructive Surgery in the Departments of Obstetrics/Gynecology/Urology, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UHCMC IRB 04-13-45; IIT #578 (Other: Allergan INC)
Record Dates: First submitted 2014-06-09; First posted 2014-06-25 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Myofascial Pain Syndromes; Myofascial Trigger Point Pain; Trigger Point Pain, Myofascial
Keywords: Myofascial Pain Syndromes; Pelvic pain; Trigger points + injections; Myofascial Trigger Point Pain; Trigger Point Pain, Myofascial; Botulinum Toxins, Type A; Botulinum Neurotoxin A; Botulinum Toxin Type A; Clostridium botulinum A Toxin; Clostridium Botulinum Toxin Type A; Oculinum
MeSH Terms: conditions — Myofascial Pain Syndromes; Pelvic Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Active Comparator): 20 patients randomly assigned to receive 100 U onabotulinumtoxinA reconstituted in 20 ml saline sequentially injected bilaterally into the pubococcygeus, iliococcygeus, coccygeus, obturator internus, and piriformis muscles.
  Interventions: Drug: OnabotulinumtoxinA
- Placebo group (Placebo Comparator): 20 patients randomly assigned to receive 20 ml of saline bilaterally into the same pelvic floor muscles.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OnabotulinumtoxinA — comparison of OnabotulinumtoxinA with placebo
  Other Names: Botox
  Arms: Treatment Group
Drug: Placebo — comparison of placebo with investigational drug OnabotulinumtoxinA
  Arms: Placebo group

SUMMARY:
This research study because is looking at woman with symptoms of chronic pelvic pain caused by short, tight, and tender pelvic floor muscles (Myofascial Pelvic Pain syndrome). The purpose of this study is to determine whether or not injections with onabotulinumtoxinA (Botox) improve symptoms of pain and tenderness. The drug being studied, Botox is FDA approved for other uses. However, Botox is not FDA approved for the use in myofascial pelvic pain (MPP). Therefore, Botox is considered experimental or research in this study.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE: Chronic pelvic pain affects 15-20% of the female population aged 18-50 years and accounts for up to 10% of gynecologic visits each year resulting in a cost of 2.8 billion dollars annually to the health care system. It is defined as non-menstrual (non-cyclic) pain that occurs on an average of two weeks per month for at least six months' duration; localized to the anatomic pelvis, anterior abdominal wall below the umbilicus, buttocks, or lumbosacral back. Many affected patients are noted to have severely short and tight pelvic floor muscles on examination (termed MPP), resulting in pelvic floor trigger points which may cause associated pelvic symptoms, including: dyspareunia, urinary urgency and frequency, symptoms of a urinary tract infection, and pelvic discomfort or heaviness.As a result of the constant, severe pain and associated symptoms, women with chronic pelvic pain are more likely to experience a decrease in their quality of life, depression, and anxiety towards their condition. The difficulty in treating chronic pelvic pain is that the etiology can be varied and multifactorial. Frequently associated with an abnormal response to an acute injury such as a pelvic infection, traumatic birth, and endometriosis or repetitive insult like chronic constipation, chronic pelvic pain can also result from prolonged pelvic floor muscle spasm and muscular hypertonicity. Specialized examination of the pelvic floor musculature in patients with chronic pelvic pain will often reveal MPP as well as 'trigger points'.11 This pain is perpetuated as a result of modifications in the neuronal pathways which maintain a set pattern of pain sensations including increased pain sensitivity (hyperalgesia), referred pain, and even changes in tissue make-up. The treatment of MPP must therefore treat the inciting injury and modify the tissue response. The effects of onabotulinumtoxinA on painful muscle were first suggested by the effects of toxin injection in patients with migraine headache. While undergoing onabotulinumtoxinA injection for cosmetic purposes, patients also suffering from migraine headaches found symptom improvement. Further follow-up studies demonstrated a 51% complete resolution and 38% a partial response noted of migraine symptoms within in 1 to 2 hours of treatment among true migraine patients. Although the mechanism of action remains unclear, onabotulinumtoxinA is believed to act by denervating autonomic nerves, thereby altering peripheral sensory nerve function and interrupting the migraine cycle of pain. The trigeminal neurovascular theory of migraine pain suggests that onabotulinumtoxinA acts not only causing muscle paralysis, but also inhibiting the transmission of any vesicles from the synaptic junction, including vasoactive intestinal peptide. This blockage of any neuromuscular junction transmission inhibits any muscle activity or efferent pain signals. Interestingly, though muscle paralysis takes about one week to manifest, pain relief occurs in 1 to 2 hours and although flaccid paralysis last for approximately 3 months, benefits for migraine pain last much longer.

STUDY RATIONALE: In MPP syndrome, prolonged muscle contraction, spasm, and inappropriately high muscle tone are thought to diminish blood supply and increase oxygen demand of the muscles of the pelvic floor. Ischemic muscle may secrete pain-producing substances, which further sensitize muscle nociceptors, alter receptor field properties, and convert wide-band mechanoreceptors to nociceptors. OnabotulinumtoxinA can directly block cholinergic neuromuscular transmission and interrupt the cascade of events that lead to hyperalgesia and allodynia. onabotulinumtoxinA plays a direct role by blocking the alpha- and gamma-motor neurons, thereby preventing the abnormal pattern of muscle contraction (eg, spasm, dystonia) that activates muscle nociceptors and sensitizes the muscle pain system through mediators.The investigators division has been utilizing pelvic floor injections of onabotulinumtoxinA as an off-label treatment for MPP in conjunction with pelvic floor physical therapy for more than 6 years. In patients with severe MPP, who often unable to tolerate any vaginal exam, or those receiving no further reduction in pelvic pain with extensive physical therapy, the investigators have been utilizing the injection of 100 U of onabotulinumtoxinA into pelvic floor trigger points with significant success. Anecdotally, treated patients report a 30-40% reduction in their pain complaints 7-10 days post-treatment which lasts for approximately 3 months. Even when the pain recurs, it is not as severe as it was pre-treatment and patients take the opportunity of the window of reduced pain to maximize further progress with pelvic floor physical therapy. Two to four weeks after pelvic floor injection, patients with severe MPP reported statistically significant changes in VAS scores before and after onabotulinumtoxinA treatment with a median reduction in VAS of -3.9 (CI for changed score -2.2, -5.6, p<0.001). Eighty percent of patients reported significant subjective improvement in their pelvic pain lasting more than 4 weeks and anecdotally lasting up to 3 to 4 months in duration. Adverse events were reported by 22% of patients and were mild, limited to: pelvic heaviness, increased pain, urinary irritation, and nausea/vomiting. However, despite these encouraging results, there is no definitive evidence that onabotulinumtoxinA is an effective treatment modality in patients with severe MPP. In their evidence-based review of the literature regarding the treatment of refractory pain with onabotulinumtoxinA, Jabbari and Machado found only level C evidence (possibly effective, may be used at discretion of clinician) when investigated the role of onabotulinumtoxinAs in the treatment of MPP. Moreover, less is known regarding the potential side effects of onabotulinumtoxinA injected into the pelvic floor muscles. Therefore, stronger randomized controlled studies are necessary to investigate the efficacy and possible side effects of pelvic floor injections of onabotulinumtoxinA in the treatment of MPP syndrome and this is actually our research proposal. It is our hope that our study will significantly change current clinical treatment protocols for MPP syndrome.

STUDY DESIGN: This is a phase I study in which participants will be randomized 1:1 (onabotulinumtoxinA:placebo), double-blinded, placebo-controlled clinical trial. Potential participants are women seeking treatment for MPP as diagnosed by the participating clinical investigators based on the following criteria: MPP is defined by at least 4 to 5 palpable trigger points on transvaginal and/or transrectal examination of the pelvic floor, which reproduces the pain for which they are seeking medical care. A trigger point is defined as an extremely tender focus of muscle causing pain radiating to other areas specific for each trigger point. A trigger point is termed 'active' if pain occurs spontaneously, and 'latent' if palpation and pressure are required to elicit pain, which may replicate symptoms or radiate to surrounding lower extremity, pelvic and abdominal sites. This study will have two arms:* Treatment group: 20 patients randomly assigned to receive 100 U onabotulinumtoxinA reconstituted in 20 ml saline sequentially injected bilaterally into the pubococcygeus, iliococcygeus, coccygeus, obturator internus, and piriformis muscles. * Placebo group: 20 patients randomly assigned to receive 20 ml of saline bilaterally into the same pelvic floor muscles. All injections will be performed using a pudendal injection tray in the clinical treatment area after obtaining consent. The patients will be randomized using a computer-generated randomization sequences in balanced blocks of four. Both the patients and physicians will be blinded to the first injection assignment. All participants with inadequate symptom control (VAS score 7 or more) at 1 months after the injection will have their treatment unblinded. Those who received placebo (saline) will be offered injection with open label onabotlulinumA. Those who previously received onabotlulinumA will not be eligible for reinjection. All patients will be followed for 6 months after the initial injection or for 6 months following the second injection. All patients who opt for a second injection will once again begin the outlined injection follow-up visit schedule.

STUDY PROCEDURES:

Screening - A detailed medical and surgical history, demographic information and review of medications will be taken from all patients suspected of having MPP. Then, a physical exam and a pelvic floor examination for myofascial trigger points will be performed. It will include an assessment of VAS at the bilateral pubococcygeus, iliococcygeus, coccygeus, obturator internus, and piriformis muscles. All VAS scores will be recorded. Post residual Void (PVR) will be recorded. Patients will have an assessment of their post residual void (PVR) and the volume will be recorded. Patients who meet inclusion criteria will be offered study participation. Patients who agree to participate will be formally consented and complete all pertinent questionnaires: * Short Form 12 (SF-12) for quality of life assessment * Patient Global Impression Index (PGI-I) for degree of bother from pelvic pain * Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ - short form 7) to assess the bladder and bowel functions * Female Sexual Function Index (FSFI) for sexual function assessment. Currently no validated questionnaire for symptoms of MPP exists.

Procedure - A pudendal block type needle is gently advanced along the outstretched fingers. Holding the needle in a near horizontal plane, the pelvic floor muscles are injected in a systematic fashion starting on the levator ani and then marching backward all the way down back to the piriformis muscle including the obturator internus muscle. The following muscles are sequentially injected with 2 cc of diluted onabotulinumtoxinA: pubococcygeus (this muscle is felt as a sling around the vagina, just proximal to the hymenal ring), iliococcygeus (palpated superiorly and laterally to pubococcygeus muscle), obturator internus (on the sidewalls of the pelvis just superior to the arcus tendineus levator ani), coccygeus (half distance between the ischial spine and sacrum), and piriformis (these muscles are palpated filling the posterolateral pelvic walls and are injected lateral to the sacrum). Careful attention is made to withdraw prior to injection to ensure no intravascular injection of the diluted onabotulinumtoxinA. Once the injection had been performed on one side of the pelvis, pressure is held for good hemostasis. The same procedure is then performed on the other side. Peri-procedural adverse events are recorded.

Post Procedure Instructions - Post treatment, all patients will be monitored for 15 minutes. Standardized post-injection instructions are given to the participant verbally and in written form. Patients will be contacted by telephone within 24-48 hours after the procedure for safety assessment. The first follow-up evaluation will be scheduled 1 month after pelvic floor injection.

Follow-Up Visits 3, 4, 5, 6, 7 & Visit 8 (Visit 8, only if Patient Received 2nd Injection) - Follow-up clinic evaluations will occur 1, 2, 3, 4 and 6 months after injection, respectively. A history will be taken and a physical examination that includes PVR assessment will be performed at each follow-up visit. VAS scores of pelvic floor muscles will be recorded. PGI-I, PFDI, PFIQ, and FSFI forms will be collected at each follow-up visit. Adverse events will be carefully monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Females age 18 years to 65 years
2. MPP for at least 6 months with pain ranked > 7/10 by VAS
3. Able to make medical decisions for herself
4. Ability to speak and understand English
5. Ability to follow study instructions and likely to complete all required visits 6 .Must give written informed consent before enrolment in this study

Exclusion Criteria:

1. Pelvic onabotulinumA injections within the last 6 months
2. Pelvic floor physical therapy (PFPT) within the last 1 months
3. Pelvic surgery within the last 1 year
4. PVR greater than 150 ml
5. Presence of interstitial cystitis/ painful bladder syndrome (IC/PBS) by the current The National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) criteria 37.
6. Evidence of pelvic pathology or other active diagnoses of acute or chronic pain syndromes including endometriosis, chronic cystitis, acute urinary tract infection, vaginitis, pelvic inflammatory disease, etc.
7. Breastfeeding, pregnant or contemplating pregnancy in the next 1 year or not on a current reliable form of birth control
8. Patients with known neurological diseases involving impaired neurotransmission, including myasthenia gravis and Charcot-Marie-Tooth disease
9. Patients who are on ambulatory anticoagulant therapy, including aspirin, who are unable to discontinue this treatment for 24 hours prior to the bladder injection
10. Women taking aminoglycosides at the time of injection (i.e. Cipro)

12. Uncontrolled clinically significant medical condition other than the condition under investigation 13. Known allergy or sensitivity to any of the components in the study medication 14. Concurrent or past (within 1 months) participation in another investigational drug or device study 15. Any condition or situation that, in the investigators opinion, may put the patients at significant risk, confound the study results, or interfere significantly with the patients participation in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
efficacy | at 1 month post treatment versus placebo
  a 30% reduction of pain and muscular spasm assessed by visual analog scale - VAS

SECONDARY OUTCOMES:
Duration of effect | 1 month post treatment versus placebo.
  Reduction of pain and muscular spasm assessed at the 1 month visit by visual analog scale - VAS
quality of life | 1 month post treatment versus placebo
  assessed by validated patient-filled questionnaires
bladder/bowel/sexual functions | 1 month post treatment versus placebo
  assessed by validated patient-filled questionnaires
complications of therapy | 1 month post treatment versus placebo
  Assessed by clinical complications of therapy (including urinary retention by PVR and other associated complaints)

OTHER OUTCOMES:
Primary Endpoint: pelvic pain scores and pelvic floor pressures | 1 month after injection
  assessed by pelvic pain scores and pelvic floor pressures
Secondary Endpoints: treatment duration effect | 1, 2, 3, 4 and 6 months after injection and/or by a change in treatment
  assessed by pelvic pain scores after injection and/or by a change in treatment
Secondary endpoint: Quality of Life | at 1, 3, and 6 months post injection
  assessed by validated patient-filled questionnaires
Secondary Endpoints: bladder/bowel functions/sexual activity | 1, 2, 3, 4 and 6 months post injection
  assessed by validated patient-filled questionnaires
Secondary Endpoints: Urinary complaints | 1, 2, 3, 4 and 6 months post injection
  assessed by urinary retention defined (PVR >150ml) and other associated complaints

CONTACTS AND LOCATIONS:
Overall Officials: Sangetta Mahajan, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (3):
- United States (3):
  - University Case Medical Center, Cleveland, Ohio
  - University Hospitals Landerbrook Health Center, Urology, Mayfield Heights, Ohio
  - University Hospitals Westlake Health Center, Urology, Westlake, Ohio